CLINICAL TRIAL: NCT02533076
Title: The Functional Consequences of the CTNS-deletion for the TRPV1-receptor in Cystinosis Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CCP13-3302-CYST
Record Dates: First submitted 2015-07-14; First posted 2015-08-26 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-07

CONDITIONS: Cystinosis
MeSH Terms: conditions — Cystinosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cystinosis Patients (Other): Cystinosis patients
  Interventions: Other: Challenge agent: capsaicin; Other: Challenge agent: placebo; Device: Mechanical stimulation with Von Frey filaments; Device: Temperature sensitivity measurement with Advanced Thermal Stimulation
- Healthy volunteers (Other): Healthy volunteers
  Interventions: Other: Challenge agent: capsaicin; Other: Challenge agent: placebo; Device: Mechanical stimulation with Von Frey filaments; Device: Temperature sensitivity measurement with Advanced Thermal Stimulation

INTERVENTIONS:
Other: Challenge agent: capsaicin — During the study period (Day 1), in each subject 3 equally spaced (minimum distance of 4 cm) 10-mm rubber O-rings (8 mm inner diameter) will be placed on the volar surface of the forearm. The most proximal ring (i.e. at least 15 cm proximal of the wrist crease) is referred to as ring number 1; the most distal ring is referred to as ring number 3; in between is ring number 2.
  In ring number 1 and 2, subjects will receive a topical dose of 1000 µg/20 µL capsaicin (single-blind). Change in dermal blood flow induced by capsaicin will be measured with Laser Doppler Imaging.
Other: Challenge agent: placebo — During the study period (Day 1), in each subject 3 equally spaced (minimum distance of 4 cm) 10-mm rubber O-rings (8 mm inner diameter) will be placed on the volar surface of the forearm. The most proximal ring (i.e. at least 15 cm proximal of the wrist crease) is referred to as ring number 1; the most distal ring is referred to as ring number 3; in between is ring number 2.
  In ring number 3, subjects will receive a topical dose of placebo (single-blind).Change in dermal blood flow induced by placebo will be measured with Laser Doppler Imaging.
Device: Mechanical stimulation with Von Frey filaments — Von Frey filaments will be used to measured the mechanical detection and pain threshold of the volunteers. The Von Frey filaments will be applied on the upper capsaicin spot in sequential order. The subject will be asked to indicate when he feels the application of the Von Frey filaments and when it hurts.
Device: Temperature sensitivity measurement with Advanced Thermal Stimulation — Temperature sensitivity (detection and pain threshold) will be determined using Advanced Thermal stimulation. A thermode will be attached to the hand of the volunteer with a baseline temperature of 32°C. The thermode will heat up and cool down with a rate of 1°C/second and the volunteer will be asked to click on a computer mouse when he feels the change in temperature and when it hurts.

SUMMARY:
Cystinosis is a rare autosomal recessive disorder, characterized by the abnormal accumulation of cystine in the lysosomes. Cystinosis is mostly caused by mutations in the cystinosin gene (CTNS). The major mutation, which is present in almost 50% of the cystinosis patients, is a 57-kb deletion. This deletion removes the first 9 exons and a part of exon 10 of the CTNS gene. Exon 10 of the CTNS gene is a upstream 5' region that encodes for the CARKL gene and also for the first two noncoding exons of the transient receptor potential channel, vanilloid subfamily member 1 (TRPV1) gene.

TRPV1 belongs to the transient receptor potential (TRP) superfamily of cation channels. TRPV1 is primarily expressed in sensory nerves and is activated by heating (>43°C) and a wide range of chemical stimuli. One of these chemical stimuli is capsaicin, the pungent ingredient in hot chilli peppers. The effect of binding of the exogenous ligand capsaicin with the TRPV1 receptor is well known to provoke the release of a number of bioactive substances including calcitonin gene-related peptide (CGRP). These substances, in turn, act on target cells in the surrounding tissue such as mast cells, immune cells and vascular smooth muscle cells. The resulting response is characterized by redness and warmth (secondary to vasodilatation), swelling (secondary to plasma extravasation) and allodynia (i.e. hypersensitivity to heat and touch secondary to alterations in the excitability of primary sensory neurons).

The present study wants to test the following hypotheses:

(i) The DBF response to topical applied capsaicin is decreased in cystinosis patients, compared to matched control subjects.

(ii) The skin sensitivity response after topical applied capsaicin is decreased in cystinosis patients, compared to matched control subjects.

(iii) The temperature sensitivity is decreased in cystinosis patients, compared to matched control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Only healthy controls: Subject is in good health, based on medical history and physical examination
* White (Caucasian) male or female subjects, aged > or = 8 year.
* Subject is capable and willing to give informed consent.

Exclusion Criteria:

* Any abnormality of the skin which may interfere with the study assessments.
* Excessive hair growth on the volar surface of the forearm.
* Excessive tanning (any exposure to sunlight or a tanning bed which would cause a sunburn reaction) throughout the study and incapable to cover the forearms for 24 hours prior to the study period.
* Subject using topical treatments on the forearm.
* History of sensitivity to the fruits of capsicum plants (e.g. chilli peppers).
* Any situation that can compromise the study, including a predictable lack of cooperation from the volunteer.
* Female subject is pregnant or breastfeeding.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the dermal blood flow response to topical applied capsaicin at 10, 20, 30, 40, 50 and 60 minutes, measured with Laser Doppler Imaging and expressed in % change to baseline | Day 1 at baseline and 10, 20, 30, 40, 50 and 60 minutes after capsaicin application
  At baseline and every 10 minutes during 60 minutes after capsaicin application. DBF measurement will be done using a Laser Doppler scanner (PIM III Perimed).

SECONDARY OUTCOMES:
Change from baseline of the skin sensitivity response after topical applied capsaicin at 10, 20, 30, 40, 50 and 60 minutes, measured with the Numerical rating scale and skin sensitivity to mechanical stimulation, measured with Von Frey filaments. | Day 1 at baseline and 10, 20, 30, 40, 50 and 60 minutes after capsaicin application
  At baseline and every 10 minutes during 60 minutes after capsaicin application, skin sensitivity to capsaicin will be measured using the Numerical rating scale (NRS) -11. Skin sensitivity to mechanical stimulation will be tested using Von Frey filaments after DBF measurements are performed.
Temperature sensitivity (detection and pain threshold), measured with Advanced Thermal stimulation and expressed in degrees Celsius. | Day 1
  Temperature sensitivity will be measured using Advanced Thermal stimulation (ATS) ( Pathway ATS Medoc) after DBF measurements are performed. A thermode will be attached to the hand of the volunteer with a baseline temperature of 32°C. The thermode will heat up and cool down with 1°C/second and the volunteers will be asked to click on a computer mouse when he/she detects the change in temperature and when it hurts.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Clinical Pharmacology, UZ Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] Buntinx L, Voets T, Morlion B, Vangeel L, Janssen M, Cornelissen E, Vriens J, de Hoon J, Levtchenko E. TRPV1 dysfunction in cystinosis patients harboring the homozygous 57 kb deletion. Sci Rep. 2016 Oct 13;6:35395. doi: 10.1038/srep35395. PMID 27734949